CLINICAL TRIAL: NCT05904353
Title: Collaboration to Improve Bone Health
Brief Title: A Study to Improve the Collaboration Between Primary and Secondary Health Care on the Treatment of Osteoporosis After a Hip Fracture.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Jakob Vangen Nordbø, Principal Investigator, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2022_35
Record Dates: First submitted 2023-05-05; First posted 2023-06-15 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Hip Fractures; Osteoporosis; Zoledronic Acid; Ambulant Nurse; Case Manager
MeSH Terms: conditions — Hip Fractures; Osteoporosis

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cluster randomized intervention regions (Experimental): Patients from the intervention regions will be followed the protocol of ambulant nurse-assisted administration of zoledronic acid
  Interventions: Procedure: Ambulant nurse-assisted administration of zoledronic acid
- Cluster randomized control regions (Active Comparator): Patients from the control regions are followed as usual. General practitioners are requested to take care of the follow-up, through the patients and the discharge summary, with annual infusions of zoledronic acid.
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: Ambulant nurse-assisted administration of zoledronic acid — Patients from the intervention regions will be followed by the protocol of ambulant nurse-assisted administration of zoledronic acid.
  Arms: Cluster randomized intervention regions
Procedure: Usual care — General practitioners are requested to take care of the follow-up, through the patients and the discharge summary, with annual infusions of zoledronic acid.
  Arms: Cluster randomized control regions

SUMMARY:
This is a study to improve the collaboration between primary and secondary health care on the treatment of osteoporosis after a hip fracture. In Akershus University Hospital, patients 75 years or older with a hip fracture, are offered treatment with an infusion of zoledronic acid 5mg, combined with vitamin D and calcium supplements, to prevent new fractures. General practitioners (GPs) are requested to take care of the follow-up on this treatment with annual infusions of zoledronic acid for 3 years.

In the opinion of the investigators, it is expedient, safe, and sensible for parts of the subsequent treatment to be provided by GPs. If hospitals take responsibility for initiating the treatment, the investigators believe that most of the subsequent monitoring and continuance of treatment can be conducted by the primary healthcare service. Despite this, the investigators suspect that many patients do not get their annual infusions of zoledronic acid after discharge from the hospital.

This quality assurance study aims to test a new system where ambulant nurses from the hospital support the GP in treating osteoporosis with the administration of zoledronic acid in the following 3 years after femoral neck fractures. Through the project, the investigators will create procedures for the administration and follow-up of zoledronic acid fitted in the setting of the GP office.

The design is a cluster randomized controlled study (RCT) where the regions are prospectively randomized to either intervention or control regions. Patients ≥ 75 years, which suffer a femoral neck fracture, are identified in our Department of Orthopedic Surgery, where they are provided the first infusion of zoledronic acid 5 mg and proposed participation in the study. Patients from the intervention regions will be followed by the protocol of ambulant nurse-assisted administration of zoledronic acid. Patients from the control regions are offered the usual care. Both patients from the control and intervention regions are asked to fill out a questionnaire after 1 year. The questionnaire will ask if the patient has got zoledronic acid as encouraged in the medical journal after discharge from the hospital. The primary study outcome is if the patients are offered treatment at a one-year follow-up or not.

Sample size calculation estimates a total sample of 130 patients based on a minimal clinically important difference of 20% follow-up between the groups. Because of high mortality, the investigators estimate the need for 200 patients.

The investigators hypothesize that the one-year follow-up is better in the intervention group than in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients 75 years or older with a hip fracture

Exclusion Criteria:

* Refuse treatment
* Another treatment of osteoporosis is indicated
* Guest patient, do not live in the admission area
* Dementia

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants offered treatment after one year | One year
  The primary study outcome is the number of participants offered treatment with zoledronic acid after one-year.

CONTACTS AND LOCATIONS:
Overall Officials: Lene Gjelseth Dalbak, MD, PHD, Study Chair — University Hospital, Akershus; Jakob Vangen Nordbø, MD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Orthopedic Department, Akershus University Hospital, Lørenskog, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No